CLINICAL TRIAL: NCT04721314
Title: Personalized Pacing: A New Paradigm for Patients With Diastolic Dysfunction or Heart Failure With Preserved Ejection Fraction
Acronym: myPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Margaret Infeld, Physician, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00000090
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Pacemaker; Diastolic Dysfunction; Diastolic Heart Failure
Keywords: Heart failure with preserved ejection fraction; Diastolic dysfunction; Resting heart rate; Personalized; Lower rate setting
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Intervention Model Description: Patients are randomized to either a personalized pacemaker lower heart rate setting based on a resting heart rate algorithm or to the conventional pacemaker lower rate setting of 60bpm.
Who Masked: Participant, Investigator
Masking Description: All investigators are blinded to patient randomization. To assess subject blinding, participants are asked at 1 month and 12 month follow up if they believed that their pacemaker lower rate was changed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Lower rate set to a higher, personalized backup heart rate (myPACE) (Experimental): Patients randomized to this group will have their pacemaker lower heart rate setting programmed to a personalized lower rate based on a resting heart rate algorithm.
  Interventions: Device: Adjustment of lower rate limit
- Lower rate left at 60 beats-per-minute (Active Comparator): Patients randomized to this group will have their pacemaker lower heart rate setting left at or programmed to the conventional pacemaker lower rate setting of 60bpm.
  Interventions: Device: Maintenance of lower rate limit

INTERVENTIONS:
Device: Adjustment of lower rate limit — Patients with preserved ejection fraction (EF >50%) and implanted pacemakers will have the lower rate limit adjusted to a personalized heart rate based on a heart rate algorithm.
  Arms: Lower rate set to a higher, personalized backup heart rate (myPACE)
Device: Maintenance of lower rate limit — Lower rate limit will be maintained at 60 beats-per-minute
  Arms: Lower rate left at 60 beats-per-minute

SUMMARY:
Recent exploratory studies suggest that pacemaker patients with diastolic dysfunction (DD) or heart failure with preserved ejection fraction (HFpEF) may benefit from a higher backup heart rate (HR) setting than the factory setting of 60 beats per minute (bpm). In this prospective double-blinded randomized controlled study, pacemaker patients with DD or overt HFpEF and either 1) intrinsic ventricular conduction or 2) conduction system or biventricular pacing will be enrolled and randomized to either a personalized lower HR setting (myPACE group, based on a height-based HR algorithm) or to the standard 60bpm backup setting (control group) for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Implanted pacemaker with either 1) intrinsic ventricular conduction or 2) conduction system or biventricular pacing or 3) RV pacing <2% and paced QRS duration <150ms
* Clinical evidence of heart failure with preserved ejection fraction or diastolic dysfunction, based on:

  * dyspnea with exertion
  * or NYHA Class ≥ II heart failure
  * or pulmonary edema on prior chest imaging or documented on exam
  * or is taking loop diuretics for heart failure
  * or had NTproBNP >400 ng/ml in the last 24 months
  * or a heart failure hospitalization in the last 2 years
  * or has diastolic dysfunction on echo
  * or has left ventricular hypertrophy on echo
  * or has left atrial (LA) dilation (LA volume/BSA index >28ml/m2)

Exclusion Criteria:

* Left ventricular ejection fraction < 50%
* Life expectancy < 12 months
* Symptomatic pulmonary disease on home oxygen
* Uncontrolled hypertension as defined by blood pressure >160/100 mmHg on two checks ≥15 minutes apart
* Hypertrophic cardiomyopathy
* More than moderate valvular disease
* Aortic valve replacement < 1 year
* Angina pectoris
* Creatinine > 2
* Hemoglobin < 8 g/dL
* Participation in another clinical trial or registry study
* Inability to follow up for regularly scheduled pacemaker appointments or to follow up for this study
* Pregnant patients or patients of childbearing age without reliable contraceptive agent (intra-uterine device, birth control implant, compliance with contraception injections or contraception pills) for the duration of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire Score | Baseline, 1 month, and 12 months
  Change in score from baseline (at enrollment) to 1 month and 12 months after enrollment.

SECONDARY OUTCOMES:
NTproBNP | Baseline, 1 month
  Change in NTproBNP level from baseline to 1 month
Hospitalization or invasive outpatient intervention for heart failure | At 12 months
Atrial Arrhythmia Burden | At 12 months
  On pacemaker reports
Loop diuretic initiation or up-titration | At 12 months
Anti-arrhythmic initiation or up-titration | At 12 months
Pacemaker-detected activity levels | At 12 months
hospitalizations or invasive outpatient intervention for heart failure exacerbation, atrial tachyarrhythmias, cerebrovascular accident, or myocardial infarction | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Meyer, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Infeld M, Cyr J, Novelli AE, Rawlings R, Wahlberg K, Plante TB, de Lavallaz JDF, Habel N, Lustgarten DL, Meyer M. Clinical Outcomes With Personalized Accelerated Physiologic Pacing in Heart Failure With Preserved Ejection Fraction: Follow-up of the myPACE Trial. JAMA Cardiol. 2025 Oct 1;10(10):1010-1015. doi: 10.1001/jamacardio.2025.2827. PMID 40864451
- [Derived] Infeld M, Wahlberg K, Cicero J, Plante TB, Meagher S, Novelli A, Habel N, Krishnan AM, Silverman DN, LeWinter MM, Lustgarten DL, Meyer M. Effect of Personalized Accelerated Pacing on Quality of Life, Physical Activity, and Atrial Fibrillation in Patients With Preclinical and Overt Heart Failure With Preserved Ejection Fraction: The myPACE Randomized Clinical Trial. JAMA Cardiol. 2023 Mar 1;8(3):213-221. doi: 10.1001/jamacardio.2022.5320. PMID 36723919